CLINICAL TRIAL: NCT02979197
Title: A Prospective Randomized Placebo Controlled Study to Evaluate the Effect of Celecoxib on the Efficacy and Safety of Amlodipine on Renal and Vascular Function in Subjects With Existing Hypertension Requiring Antihypertensive Therapy
Brief Title: Evaluation of Celecoxib Effects on Amlodipine in Subjects With Existing Hypertension Requiring Antihypertensives
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kitov Pharma Ltd (Unknown)
Responsible Party: Sponsor
Organization: KitovPharma (Unknown)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: KIT-302-03-02; 2016-002214-47 (EudraCT Number)
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Hypertension
Keywords: High blood pressure; Systolic blood pressure; Diastolic blood pressure; Antihypertensive
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Amlodipine+Celecoxib (Experimental): OE 10 mg amlodipine besylate tablet + OE 200 mg celecoxib capsule qd for 14 days
  Interventions: Drug: OE 10 mg amlodipine besylate tablet; Drug: OE 200 mg celecoxib capsule
- Amlodipine+Placebo (Active Comparator): OE 10 mg amlodipine besylate tablet + matched placebo for OE celecoxib capsule qd for 14 days
  Interventions: Drug: OE 10 mg amlodipine besylate tablet; Drug: Matched placebo for OE celecoxib capsule
- Placebo+Placebo (Sham Comparator): Matched placebo for OE amlodipine besylate tablet + matched placebo for OE celecoxib capsule qd for 14 days
  Interventions: Drug: Matched placebo for OE amlodipine besylate tablet; Drug: Matched placebo for OE celecoxib capsule

INTERVENTIONS:
Drug: OE 10 mg amlodipine besylate tablet
  Other Names: OE 10 mg Norvasc tablet
  Arms: Amlodipine+Celecoxib; Amlodipine+Placebo
Drug: OE 200 mg celecoxib capsule
  Other Names: OE 200 mg Celebrex capsule
  Arms: Amlodipine+Celecoxib
Drug: Matched placebo for OE amlodipine besylate tablet
  Other Names: Matched placebo for OE Norvasc tablet
  Arms: Placebo+Placebo
Drug: Matched placebo for OE celecoxib capsule
  Other Names: Matched placebo for OE Celebrex capsule
  Arms: Amlodipine+Placebo; Placebo+Placebo

SUMMARY:
The purpose of this study was to evaluate the effect of celecoxib on the efficacy and safety of amlodipine besylate on renal and vascular function in subjects with existing hypertension requiring antihypertensive therapy.

Kitov Pharma Ltd. (Kitov) is developing KIT-302, an oral fixed combination drug product (FCDP) consisting of the calcium channel blocker amlodipine besylate and the nonsteroidal anti-inflammatory drug (NSAID) celecoxib, as a "convenience reformulation" FCDP to facilitate and improve patient compliance with the once a day (qd) administration of its individual components, amlodipine and celecoxib.

The formulation of KIT-302 consists of amlodipine besylate and celecoxib co-formulated in a single immediate release tablet. However, for this study (KIT-302-03-02), commercial celecoxib capsules (Celebrex®) and commercial amlodipine besylate tablets (Norvasc®) were separately over-encapsulated (OE) and matched placebos were used to allow for blinding.

Kitov completed a phase 3 pivotal trial in subjects with newly diagnosed hypertension (KIT-302-03-01) demonstrating that the amlodipine + celecoxib combination was statistically non-inferior to amlodipine monotherapy with regard to reduction of blood pressure. Further, trends towards superior blood pressure lowering effects and improved renal function were observed for the combination. This study (KIT-302-03-02) was conducted to quantify the beneficial renovascular effects noted in the prior study in subjects with existing hypertension requiring antihypertensive therapy.

On May 31, 2018, the United States (US) Food and Drug Administration (FDA) approved KIT-302, under the brand name Consensi® (amlodipine and celecoxib) tablets [New Drug Application (NDA) 210045] for the following indication: "patients for whom treatment with amlodipine for hypertension and celecoxib for osteoarthritis are appropriate. Lowering blood pressure reduces the risk of fatal and nonfatal cardiovascular events, primarily strokes and myocardial infarctions."

DETAILED DESCRIPTION:
This was a multi-center, randomized, double blind, placebo controlled study to evaluate the effect of celecoxib on the efficacy, safety, and pharmacokinetics of amlodipine in subjects with existing hypertension requiring antihypertensive therapy. Approximately 105 eligible subjects were to be randomized 3:3:1 to one of three treatment arms.

Arm 1:OE 10 mg Norvasc tablet+OE 200 mg Celebrex capsule (amlodipine+celecoxib arm)

Arm 2:OE 10 mg Norvasc tablet+matched placebo for OE Celebrex capsule (amlodipine+placebo arm)

Arm 3:Matched placebo for OE Norvasc tablet+matched placebo for OE Celebrex capsule (placebo+placebo arm).

Following an up to 14-day screening phase, eligible subjects were randomized to one of the 3 treatment arms. All drugs were to be administered orally qd for 14 days for a total of 14 doses. Visits at the clinic took place at the start and at the end of the screening phase, at Study Day 0 (start of treatment), Day 6, Day 7, Day 13 (end of treatment), Day 14 and Day 28 (end of follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Adult 40 to 75 years of age
2. Existing hypertension that is being treated using pharmacological therapy with a single agent that is not a calcium channel blocker
3. SBPday > 135 and ≤ 169 mmHg and average daytime (9:00 to 21:00) ambulatory diastolic blood pressure (DBPday) ≤ 110 mmHg at Day 0 (after the 10- to 14-day washout from prior blood pressure medication)
4. Body Mass Index of 18.5 to 34.9 kg/m2
5. Healthy (other than hypertension) as determined by the Investigator based on medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests
6. A negative pregnancy test at initial screening visit
7. If woman of childbearing potential, agree to use a highly effective form of birth control while on study (from Screening through final study visit)
8. Able to comprehend and sign an informed consent form.

Exclusion Criteria:

1. Resting SBP > 169 mmHg or a resting DBP > 110 mmHg at initial screening visit while on their standard antihypertensive therapy (where resting is defined as supine for at least 10 minutes with minimal interaction)
2. Weight < 55 kg
3. Fragile health
4. Evidence of clinically significant findings on screening evaluations (clinical, laboratory, and ECG) which, in the opinion of the Investigator would pose a safety risk or interfere with appropriate interpretation of safety data
5. Current or recent history (within four weeks prior to initial screening visit) of a clinically significant bacterial, fungal, or mycobacterial infection
6. Current clinically significant viral infection
7. History of malignancy, with the exception of cured basal cell or squamous cell carcinoma of the skin
8. Major surgery within four weeks prior to initial screening visit
9. Presence of a malabsorption syndrome possibly affecting drug absorption (e.g., Crohn's disease or chronic pancreatitis)
10. Active peptic ulceration or history of gastrointestinal bleeding
11. History of myocardial infarction, congestive heart failure, or stroke
12. Any current cardiovascular disease (other than hypertension)
13. History of psychotic disorder
14. History of alcoholism or drug addiction or current alcohol or drug use that, in the opinion of the Investigator, will interfere with the subject's ability to comply with the dosing schedule and study evaluations
15. History of any illicit drug use within one year prior to initial screening visit
16. Positive drug screen at initial screening visit. A positive drug screen for opiates only (with all other drug tests negative) will not be a basis for exclusion if the subject took over-the-counter narcotics as indicated on the product label within 24 hours prior to the drug screen
17. Current treatment or treatment within 30 days prior to first dose of study drugs with another investigational drug or current enrollment in another clinical trial
18. Known history of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
19. Known hypersensitivity to amlodipine or celecoxib
20. Known hypersensitivity to the inactive ingredients in the over-encapsulated (OE) study drugs
21. Asthma, acute rhinitis, nasal polyps, angioneurotic oedema, urticaria or other allergic type reactions after taking acetylsalicylic acid or NSAIDs including cyclooxygenase-2 inhibitors
22. Subjects who, in the opinion of the Investigator, are unable or unlikely to comply with the dosing schedule and study evaluations
23. Pregnant or lactating
24. Unable to correctly use ambulatory blood pressure monitor after instruction on its use
25. Subjects with Child-Pugh Class B or C cirrhosis
26. Subjects currently taking a calcium channel blocker or any NSAID for any reason will be excluded. Subjects will not be withdrawn from these drugs to be enrolled in the trial
27. Subjects that took a calcium channel blocker in the past for any indication
28. Creatinine clearance < 50 ml/min as estimated by the Cockroft-Gault equation
29. Known cytochrome P450 2C9 poor metabolizer
30. Subjects with allergy or hypersensitivity to sulfonamides

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Paul Waymack, MD, PhD, Study Director — Kitov Pharma Ltd
Locations (9):
- United Kingdom (9):
  - Oldfield Surgery, Bath
  - Celerion, Belfast
  - Hathaway Medical Centre, Chippenham
  - Rowden Surgery, Chippenham
  - Barts Health NHS Trust, Barts Queen Mary University of London, William Harvey Heart Centre, London
  - Medicines Evaluation Unit Ltd., Manchester
  - St Chad's Surgery, Radstock
  - Bradford Road Medical Centre, Trowbridge
  - Adcroft Surgery, Trowbridge

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligibility assessments were made at Initial Screening (Day -14 to -10), Final Screening (Day -1), and prior to randomization (Day 0). Subjects who met eligibility criteria at Initial Screening underwent a 10- to 14-day washout from their blood pressure medication and those who continued to meet criteria at the end of the washout were randomized.
Period: Overall Study
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Placebo
Started | 48 | 49 | 8
Completed | 44 | 45 | 8
Not Completed | 4 | 4 | 0
Not completed — Adverse Event | 4 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Subject unable to commit to study dates | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Placebo | Total
Number analyzed (Participants) | 48 | 49 | 8 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (7.13) | 56.7 (7.43) | 52.5 (7.84) | 55.8 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 4 | 39
  Male | 31 | 31 | 4 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 46 | 47 | 7 | 100
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 48 | 49 | 8 | 105
SBPday [Mean (Standard Deviation); unit: mmHg] — Average daytime (9:00 to 21:00) ambulatory systolic blood pressure measured at Day -1
  mmHg | 148.0 (7.95) | 150.0 (8.25) | 151.5 (10.91) | 149.2 (8.33)

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Daytime (9:00 to 21:00) Ambulatory Systolic Blood Pressure (SBPday)
Description: An ambulatory blood pressure monitor (ABPM) fitted to upper arm was used for continuous recording of blood pressure over three 25-hour periods: Days -1 to 0 (Baseline), Days 6 to 7, & Days 13 to 14. The ABPM recorded blood pressure every 20 minutes between 09:00 and 21:59 and every 30 minutes between 22:00 and 08:59. SBPday was calculated by averaging all of the systolic blood pressure measurements between the protocol-defined first & last study measurements of the period that fell between 9:00 and 21:00; measurements during the first hour (white-coat window) were not included. Change in SBPday was calculated by subtracting the Baseline value from the end of study value (Day 13 to Day 14 period). If the Day 13 to Day 14 value was not available, the Day 6 to Day 7 value was used [last observation carried forward (LOCF) method]. A negative value for change in SBPday indicates a decrease in systolic blood pressure and a positive value indicates an increase.
Time Frame: Baseline and 14 days
Population: Intent-to-treat (ITT) population = all randomized subjects with a valid Baseline (Day -1 to Day 0) ABPM measurement. The primary endpoint of this trial was a comparison of the mean change in SBPday between the amlodipine+celecoxib and amlodipine+placebo arms (non-inferiority trial). Comparison to placebo+placebo was not part of primary endpoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo
Number analyzed (Participants) | 48 | 48
mmHg | -8.0 (8.24) | -9.8 (8.89)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; LOCF method was used. Primary efficacy analysis was based on the difference between the Amlodipine+Celecoxib and Amlodipine+Placebo (arms 1 and 2, respectively) in the mean change in SBPday from Baseline to final (Day 13), where a subject completed the 14-day treatment plan, or to Day 6, where a subject was withdrawn from treatment before the Day 13 dose but after the Day 6 dose, or to baseline, where a subject was withdrawn before the Day 6 dose; Test type: Non-Inferiority — A two-sample t-test was used to test the one-sided hypothesis that treatment with Amlodipine+Celecoxib (arm 1) was non-inferior to half of the effect achieved with Amlodipine+Placebo (arm 2). The primary efficacy endpoint was considered met if the lower limits of the 97.5% one-side confidence interval (CI) for the difference in SBPday change in arm 1 and 50% of the mean change in arm 2 was less than 0; p = 0.024, t-test, 2 sided

2. Secondary Outcome: Change in Body Weight
Description: Body weight was measured at the Initial Screening Visit (Day -10 to -14), at Baseline (Day 0), and at Days 7 and 14. The measurements were made using a calibrated scale with the subject wearing underwear and a light gown. Change in body weight was calculated by subtracting the Baseline value from the end of treatment value (recorded on Day 14). If the Day 14 value was not available, the Day 7 value was used (LOCF method). A negative value for change in body weight indicates a decrease in body weight and a positive value indicates an increase.
Time Frame: Baseline and 14 days
Population: ITT population [i.e., all randomized subjects with a valid Baseline (Day -1 to Day 0) ABPM measurement]. A secondary endpoint of this trial was a comparison of the mean change in body weight between all three treatment arms [analysis of variance (ANOVA) F test]. Thus, mean values for all three arms are presented.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Placebo
Number analyzed (Participants) | 48 | 48 | 8
kg | 0.3 (1.02) | -0.3 (1.03) | -1.5 (3.95)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo vs Placebo+Placebo; A serial gatekeeping strategy was used for secondary efficacy analyses. If, and only if, statistical significance was achieved for the primary endpoint (SBPday), a secondary hierarchical analysis was to be used to evaluate secondary efficacy endpoints and was only to proceed from one to the next if the alpha was met for the prior; if the alpha was not met, analysis was performed for informational purposes only. Mean change in body weight was the 1st of the four secondary efficacy endpoints; Test type: Other — ANOVA F-test was used to compare the mean changes in body weight from baseline to end of treatment among the three treatment arms. The omni-bus test was to conclude if any differences existed; p = 0.006, ANOVA

3. Secondary Outcome: Change in Average 24-hour Ambulatory Systolic Blood Pressure (SBP24h)
Description: An ABPM fitted to upper arm was used for continuous recording of blood pressure over three 25-hour periods: Days -1 to 0 (Baseline), Days 6 to 7, & Days 13 to 14. The ABPM recorded blood pressure every 20 minutes between 09:00 and 21:59 and every 30 minutes between 22:00 and 08:59. SBP24h was calculated by averaging all of the systolic blood pressure measurements between the protocol-defined first & last study measurements of the period; measurements during the first hour (white-coat window) were not included. Change in SBP24h was calculated by subtracting the Baseline value from the end of study value (Day 13 to Day 14 period). If the Day 13 to Day 14 value was not available, the Day 6 to Day 7 value was used (LOCF method). A negative value for change in SBP24h indicates a decrease in systolic blood pressure and a positive value indicates an increase.
Time Frame: Baseline and 14 days
Population: ITT population [i.e., all randomized subjects with a valid Baseline (Day -1 to Day 0) ABPM measurement]. A secondary endpoint of this trial was the comparison of the mean change in SBP24h between the amlodipine+celecoxib and amlodipine+placebo arms (superiority trial). Comparison to placebo+placebo was not part of this endpoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo
Number analyzed (Participants) | 48 | 48
mmHg | -8.2 (7.80) | -8.5 (8.47)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; A serial gatekeeping strategy was used for secondary efficacy analyses. If, and only if, statistical significance was achieved for the primary endpoint (SBPday), a secondary hierarchical analysis was to be used to evaluate secondary efficacy endpoints and was only to proceed from one to the next if the alpha was met for the prior; if the alpha was not met, analysis was performed for informational purposes only. Mean change in SBP24h was the 2nd of the four secondary efficacy endpoints; Test type: Superiority — A two-sample t-test for superiority was used to test the one-sided hypothesis that treatment with Amlodipine+Celecoxib lowered SBP24h to a greater degree than Amlodipine+Placebo; p = 0.826, t-test, 2 sided

4. Secondary Outcome: Change in Average 24-hour Ambulatory Diastolic Blood Pressure (DBP24h)
Description: An ABPM fitted to upper arm was used for continuous recording of blood pressure over three 25-hour periods: Days -1 to 0 (Baseline), Days 6 to 7, & Days 13 to 14. The ABPM recorded blood pressure every 20 minutes between 09:00 and 21:59 and every 30 minutes between 22:00 and 08:59. DBP24h was calculated by averaging all of the diastolic blood pressure measurements between the protocol-defined first & last study measurements of the period; measurements during the first hour (white-coat window) were not included. Change in DBP24h was calculated by subtracting the Baseline value from the end of study value (Day 13 to Day 14 period). If the Day 13 to Day 14 value was not available, the Day 6 to Day 7 value was used (LOCF method). A negative value for change in DBP24h indicates a decrease in diastolic blood pressure and a positive value indicates an increase.
Time Frame: Baseline and 14 days
Population: ITT population [i.e., all randomized subjects with a valid Baseline (Day -1 to Day 0) ABPM measurement]. A secondary endpoint of this trial was the comparison of the mean change in DBP24h between the amlodipine+celecoxib and amlodipine+placebo arms (superiority trial). Comparison to placebo+placebo was not part of this endpoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo
Number analyzed (Participants) | 48 | 48
mmHg | -4.4 (4.68) | -3.8 (5.27)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; A serial gatekeeping strategy was used for secondary efficacy analyses. If, and only if, statistical significance was achieved for the primary endpoint (SBPday), a secondary hierarchical analysis was to be used to evaluate secondary efficacy endpoints and was only to proceed from one to the next if the alpha was met for the prior; if the alpha was not met, analysis was performed for informational purposes only. Mean change in DBP24h was the 3rd of the 4 secondary efficacy endpoints; Test type: Superiority — A two-sample t-test for superiority was used to test the one-sided hypothesis that treatment with Amlodipine+Celecoxib lowered DBP24h to a greater degree than Amlodipine+Placebo; p = 0.500, t-test, 2 sided

5. Secondary Outcome: Change in Creatinine Clearance
Description: Subjects had blood collected for the measurement of creatinine at the Initial Screening Visit (Day -10 to -14), at Baseline (Day 0), and at Days 7 and 14. Estimated creatinine clearance was calculated using Cockcroft-Gault equation: (140 - age) X body weight (kg)/72 X serum creatinine concentration (mg/dL); multiplied by 0.85 for women. Change in creatinine clearance was calculated by subtracting the Baseline value from the end of treatment value (recorded on Day 14). If the Day 14 value was not available, the Day 7 value was used (LOCF method). A negative value for change in creatinine clearance indicates a decrease in creatinine clearance and a positive value indicates an increase.
Time Frame: Baseline and 14 days
Population: ITT population [i.e., all randomized subjects with a valid Baseline (Day -1 to Day 0) ABPM measurement]. A secondary endpoint of this trial was the comparison of the mean change in creatinine clearance between the amlodipine+celecoxib and amlodipine+placebo arms (superiority trial). Comparison to placebo+placebo was not part of this endpoint.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo
Number analyzed (Participants) | 48 | 48
mL/min | 4.9 (10.62) | 3.4 (20.96)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; A serial gatekeeping strategy was used for secondary efficacy analyses. If, and only if, statistical significance was achieved for the primary endpoint (SBPday), a secondary hierarchical analysis was to be used to evaluate secondary efficacy endpoints and was only to proceed from one to the next if the alpha was met for the prior; if the alpha was not met, analysis was performed for informational purposes only. Mean change in creatinine clearance was the 4th of 4 secondary efficacy endpoints; Test type: Superiority — A two-sample t-test for superiority was used to test the one-sided hypothesis that treatment with Amlodipine+Celecoxib improved creatinine clearance to a greater degree than Amlodipine+Placebo; p = 0.668, t-test, 2 sided

6. Secondary Outcome: Occurrence of Treatment Emergent Adverse Events
Description: Treatment emergent adverse events (TEAEs) included any untoward medical occurrence that initiated or worsened after the first dose of study drugs and within 14 days of the last dose of study drugs.
Time Frame: 1 month
Population: Safety population = all randomized subjects who received at least one dose of study drug. The occurrence of TEAEs was compared between all three arms (Chi-square test), as well as between the amlodipine+celecoxib and amlodipine+placebo arms (exact logistic regression model). Comparison to placebo+placebo was not part of this latter analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Placebo
Number analyzed (Participants) | 48 | 49 | 8
Participants | 35 | 32 | 6
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo vs Placebo+Placebo; Test type: Superiority — Differences in the occurrence of TEAEs between treatment arms were evaluated using Chi-square test; p = 0.675, Chi-squared; Computed on the number of subjects who had at least one TEAE
Statistical Analysis 2: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; Test type: Superiority; p = 0.555, Regression, Logistic; TEAE (1=at least one TEAE occurred for the subject; 0=otherwise) as dependent variable and treatment as fixed effect

7. Secondary Outcome: Non-transformed Plasma Concentration of Amlodipine
Description: A venous blood sample was collected 24 hours ± 1 hour after the last dose of study drugs (i.e., on Day 14). The blood sample was processed to plasma and the concentration of amlodipine measured using a validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) method. The resulting concentrations, without logarithmic transformation, were used for the comparison between the amlodipine+celecoxib and amlodipine+placebo arms to evaluate the effect of celecoxib on the mean non-transformed plasma concentrations of amlodipine.
Time Frame: 24 hours post-dose on Day 14
Population: Pharmacokinetic (PK) population = all subjects enrolled at an Investigational Site with ultraviolet- (UV-) shielded lights who had blood drawn on Day 14, 24 hours ± 1 hour after receiving the final dose of study drugs for the measurement of plasma amlodipine concentration; only treatment arms that included amlodipine were included in the analyses.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo
Number analyzed (Participants) | 23 | 20
ng/mL | 15.9 (5.72) | 18.3 (7.21)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; For this analysis, all values below the limit of quantification were treated as 0; Test type: Superiority; p = 0.226, t-test, 2 sided

8. Secondary Outcome: Log-transformed Plasma Concentration of Amlodipine
Description: A venous blood sample was collected 24 hours ± 1 hour after the last dose of study drugs (i.e., on Day 14). The blood sample was processed to plasma and the concentration of amlodipine measured using a validated LC-MS/MS method. The concentrations were logarithmically transformed and used for the comparison between the amlodipine+celecoxib and amlodipine+placebo arms to evaluate the effect of celecoxib on the mean log-transformed plasma concentrations of amlodipine.
Time Frame: 24 hours post-dose on Day 14
Population: PK population = all subjects enrolled at an Investigational Site with ultraviolet- (UV-) shielded lights who had blood drawn on Day 14, 24 hours ± 1 hour after receiving the final dose of study drugs for the measurement of plasma amlodipine concentration; only treatment arms that included amlodipine were included in the analyses.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo
Number analyzed (Participants) | 23 | 20
ng/mL | 2.7 (0.44) | 2.8 (0.36)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; For this analysis, all values below the limit of quantification (BLQ) were treated as 0.04 ng/mL. Assignment of BLQ values to a nonzero number allowed computation of the log transformation. The selection of 0.04 ng/mL was based on the lower limit of quantification of the validated bioanalytical method (0.05 ng/mL) and selecting the next lowest number at the hundredth decimal place; Test type: Superiority; p = 0.215, t-test, 2 sided

9. Other Pre Specified Outcome: Change in Serum Creatinine
Description: Subjects had blood collected for the measurement of creatinine at the Initial Screening Visit (Day -10 to -14), at Baseline (Day 0), and at Days 7 and 14. Change in serum creatinine was calculated by subtracting the Baseline value from the end of treatment value (recorded on Day 14). A negative value for change in serum creatinine indicates a decrease in creatinine and a positive value indicates an increase.
Time Frame: Baseline and 14 Days
Population: Safety population = all randomized subjects who received at least one dose of study drug
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Placebo
Number analyzed (Participants) | 48 | 49 | 8
μmol/L | -2.8 (5.56) | -2.4 (10.19) | -1.9 (4.61)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib; Renal function was analyzed by evaluating the decreases in serum creatinine from baseline to Day 14 for each treatment arm and between treatment arms by ANCOVA. This analysis was for the Amlodipine+Celecoxib arm from baseline to Day 14; Test type: Superiority; p = 0.0005, ANCOVA; Adjusted mean = -3.48 μmol/L; 95% confidence interval = -5.4 to -1.6
Statistical Analysis 2: Comparison: Amlodipine+Placebo; Renal function was analyzed by evaluating the decreases in serum creatinine from baseline to Day 14 for each treatment arm and between treatment arms by ANCOVA. This analysis was for the Amlodipine+Placebo arm from baseline to Day 14; Test type: Superiority; p = 0.0750, ANCOVA; Adjusted mean = -1.72 μmol/L; 95% confidence interval = -3.6 to 0.2
Statistical Analysis 3: Comparison: Placebo+Placebo; Renal function was analyzed by evaluating the decreases in serum creatinine from baseline to Day 14 for each treatment arm and between treatment arms by ANCOVA. This analysis was for the Placebo+Placebo arm from baseline to Day 14; Test type: Superiority; p = 0.4184, ANCOVA; Adjusted mean = -1.92 μmol/L; 95% confidence interval = -6.6 to 2.8
Statistical Analysis 4: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; Renal function was analyzed by evaluating the decreases in serum creatinine from baseline to Day 14 for each treatment arm and between treatment arms by ANCOVA. This analysis was for the comparison between the Amlodipine+Celecoxib and Amlodipine+Placebo arms; Test type: Superiority; p = 0.2022, ANCOVA; Adjusted mean = -1.76 μmol/L; 95% confidence interval = -4.5 to 1.0
Statistical Analysis 5: Comparison: Amlodipine+Celecoxib vs Placebo+Placebo; Renal function was analyzed by evaluating the decreases in serum creatinine from baseline to Day 14 for each treatment arm and between treatment arms by ANCOVA. This analysis was for the comparison between the Amlodipine+Celecoxib and Placebo+Placebo arms; Test type: Superiority; p = 0.5410, ANCOVA; Adjusted mean = -1.56 μmol/L; 95% confidence interval = -6.6 to 3.5
Statistical Analysis 6: Comparison: Amlodipine+Placebo vs Placebo+Placebo; Renal function was analyzed by evaluating the decreases in serum creatinine from baseline to Day 14 for each treatment arm and between treatment arms by ANCOVA. This analysis was for the comparison between the Amlodipine+Placebo and Placebo+Placebo arms; Test type: Superiority; p = 0.9397, ANCOVA; Adjusted mean = 0.19 μmol/L; 95% confidence interval = -4.9 to 5.2

ADVERSE EVENTS:
Time Frame: 1 month; TEAEs include any untoward medical occurrence that initiated or worsened after the first dose of study drugs and within 14 days of the last dose of study drugs.
Description: Subjects were instructed to report all adverse events (AEs) experienced during the study, and subjects were assessed for the occurrence of AEs throughout the study. Secondary safety assessments included physical examination, body weight, vital signs, orthostatic hypotension evaluations, 12-lead electrocardiogram, hematology, serum chemistry and urinalysis, and any clinically significant findings on these assessments were reported as AEs.
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/49 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/49 | 0/8
Other Adverse Events (participants affected / at risk) | 25/48 | 23/49 | 6/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amlodipine+Celecoxib (N=48) | Amlodipine+Placebo (N=49) | Placebo+Placebo (N=8)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 3 (6) | 0 (0)
Oedema peripheral (General disorders) | 7 (7) | 4 (5) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (2)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (8) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 10 (12) | 9 (13) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (10) | 9 (10) | 2 (3)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-12-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT02979197/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT02979197/SAP_001.pdf